CLINICAL TRIAL: NCT00992212
Title: A Phase II, Open Label Study to Evaluate the Immunogenicity, Tolerability and Safety of an Adjuvanted, Inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in Healthy Subjects Aged 18 Years and Above
Brief Title: Immunogenicity, Tolerability and Safety of One or Two Doses of an Adjuvanted Swine-origin A H1N1 Influenza Vaccine in Healthy Subjects 18 or More Years of Age Both Vaccinated and Not Yet Vaccinated Against Seasonal Influenza 2009/10
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V111_04
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2012-01

CONDITIONS: Pandemic Influenza Disease
Keywords: Pandemic influenza; vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group A (Seasonal TIV + 7.5mcg HA+ full dose MF59) (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine
- Group B (Ajuvanted Seasonal TIV + 7.5mcg HA+ full dose MF59) (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine
- Group C (7.5mcg HA+ full dose MF59) (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine
- Group D (7.5mcg HA+ full dose MF59 + Seasonal TIV) (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine
- Group E (3.75mcg HA+ ½ dose MF59+ Seasonal TIV) (Experimental)
  Interventions: Biological: Monovalent A/H1N1 influenza vaccine

INTERVENTIONS:
Biological: Monovalent A/H1N1 influenza vaccine — This trial will be performed at multiple sites; appr. 160 subjects exposed to the annual vaccine registration will be invited to take part into this study. In addition, a total of 224 healthy subjects not yet exposed to the seasonal influenza vaccines will be enrolled.

SUMMARY:
This present study, a phase II, open label study will evaluate the immunogenicity, tolerability and safety of an adjuvanted, inactivated Novel Swine Origin A/H1N1 Monovalent Subunit Influenza Virus Vaccine in healthy subjects aged 18 years and above. This study will explore the effect of the previous and concomitant exposure to a seasonal influenza vaccination to the immunogenicity and safety profile of two different doses of an adjuvanted H1N1sw vaccine.

DETAILED DESCRIPTION:
At enrolment, subjects were stratified into two age strata (18 to 60 years, over 60 years). Total duration of the study is eight weeks, which include two weeks for enrolment and 6 weeks for study participation. Vaccinations were to be administered on day 1 and day 22. Blood samples were collected at day 1 (baseline, before the first vaccination), at day 22 (before the second vaccination), at day 29 (one week after the second vaccination) and at day 43 (three weeks after the second vaccination). Sera were tested by Hemagglutination Inhibition (HI) and Microneutralization (MN) assays. Safety was assessed until 3 weeks after the first and second vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. For study Groups A and B : subjects aged 18 years and above on the day of enrollment, who took part to the seasonal trials for the 2009/10 vaccine registration; For study Groups C to E: subjects aged 18 years and above on the day of enrollment, not yet exposed to the current seasonal formulation (2009/10 for NH) of the influenza vaccines;
2. Individuals in good health as determined by medical history, physical examination and clinical judgment of the investigator;
3. Documented consent obtained after the nature of the study has been explained according to local regulatory requirements;
4. Individuals are able to comply with all study procedures and are available for all clinic visits scheduled in the study.
5. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

1. Individuals who are not able to comprehend and to follow all required study procedures; individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study;
2. Individuals with history or any illness that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study;
3. Individuals who have had received an influenza vaccine for the 2009/10 NH influenza season (for subjects to be included in Groups C to E only) prior to Visit 1;
4. Individuals who have had documented confirmed or suspected influenza disease within 6 months prior to Day 1.
5. Receipt of another investigational agent within 4 weeks prior to enrollment, or before completion of the safety follow-up period in this or in another study;
6. Individuals who received any other vaccines within 4 weeks prior to enrollment in this study and individuals who have ever received blood, blood products and/or plasma derivatives in the past 12 weeks;
7. Individuals with axillary temperature ≥ 38.0°C within 3 days of study vaccination;
8. Known or suspected impairment/alteration of immune function, for example resulting from:

   * receipt of immunosuppressive therapy,
   * cancer chemotherapy,
   * receipt of immunostimulants within 60 days prior to Visit 1,
   * receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within 3 months prior to Visit 1 or planned during the full length of the study,
   * known HIV infection or HIV-related disease.
9. Surgery planned during the study period;
10. If female, of childbearing potential, and has not used any of the "acceptable contraceptive methods" for at least 2 months prior to study entry;
11. Females who are pregnant or nursing (breastfeeding) mothers, or females of childbearing potential who are sexually active and have not used or do not plan to use acceptable birth control measures during the first 3 weeks after vaccination.
12. Members of the research staff or their relatives (research staff are individuals with direct or indirect contact with trial subjects, or study site personnel who have access to any study documents containing subject information, including: e.g. receptionists, persons scheduling appointments or making screening calls, regulatory specialists, laboratory technicians); hospital personnel and health care providers not involved in the study can be enrolled.

Min Age: 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity, safety and tolerability of 1 and 2 IM doses of MF59-H1N1sw flu vaccine in adult-elderly subjects previously exposed to 09/10 NH TIV and in those not yet vaccinated against flu season 09/10. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (5):
- Italy (5):
  - 01, Chieti
  - 05, Ferrara
  - 04, Genova
  - 02, Lanciano
  - 03, Mira 30034 Pianiga,

REFERENCES:
- [Result] Gasparini R, Schioppa F, Lattanzi M, Barone M, Casula D, Pellegrini M, Veitch K, Gaitatzis N. Impact of prior or concomitant seasonal influenza vaccination on MF59-adjuvanted H1N1v vaccine (Focetria) in adult and elderly subjects. Int J Clin Pract. 2010 Mar;64(4):432-8. doi: 10.1111/j.1742-1241.2009.02309.x. Epub 2009 Dec 17. PMID 20039974